CLINICAL TRIAL: NCT03886207
Title: Efficacy of Foot Baths With and Without Ginger Powder Additive on the Subjective Feeling of Warmth and on Body Core Temperature of Adolescents With Anorexia Nervosa - a Randomized, Controlled Pilot Study
Brief Title: Treatment Trial of Thermoregulatory Disturbances in Adolescent Anorexia Nervosa Patients With Either Ginger Powder Footbaths or Warm Water Footbaths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Filderklinik, Filderstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANS_03
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Adolescent Anorexia Nervosa
Keywords: Anorexia; Footbath; Ginger powder; Thermogenic substances; Thermoregulation; External applications; Anthroposophic medicine; Eating disorders
MeSH Terms: conditions — Anorexia; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants are age and core body temperature stratified and then randomized to one of the two groups (footbath with warm water with additional ginger powder or warm water only). Assessments are taken before and after the six-week intervention phase as well as at six-month follow-up.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm water with ginger powder footbath (Experimental): Participants who receive a warm water with added ginger powder footbath four times a week over a six-week period.
  Interventions: Other: ginger powder footbath
- Warm water only footbath (Active Comparator): Participants who receive a warm water only footbath four times a week over a six-week period.
  Interventions: Other: warm water only footbath

INTERVENTIONS:
Other: ginger powder footbath — 38-40° C warm water footbath with an additive of dried ginger powder reaching up to mid-calf level, as practiced in anthroposophic medicine
  Arms: Warm water with ginger powder footbath
Other: warm water only footbath — 38-40° C warm water footbath without any additive reaching up to mid-calf level
  Arms: Warm water only footbath

SUMMARY:
A study to explore whether warm water footbaths with added ginger powder can improve thermoregulatory processes in adolescent anorexia nervosa patients and provide them with an increase in subjective feeling of warmth. The participants will receive a warm footbath four times a week for six weeks with a physiological and psychological testing point once before the beginning of the six-week footbath period and once after.

DETAILED DESCRIPTION:
This is a two-arm randomized controlled trial to evaluate the efficacy of warm water footbaths with added ginger powder (experimental) compared to warm water only footbaths (control) in adolescent anorexia nervosa patients. Participants will receive footbaths 4 times per week before bed-time over a period of six weeks.The main focus is on subjective increase in overall body warmth. Moreover, core body temperature, skin temperature at the extremities and several psychological as well as physiological scores and parameters are assessed before and after the six-week intervention. A follow-up is planned at six months post intervention, where core body temperature, physiological and psychological parameters are once more tested.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis: Anorexia nervosa
* written informed consent of participants and legal guardians

Exclusion Criteria:

* other eating disorder diagnosis apart from Anorexia nervosa
* known allergic reaction to ginger

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Chnge in Subjective feeling of overall warmth | Baseline (pre intervention), 6 weeks after baseline (post intervention)
  Self-reported feeling of overall warmth measured using the HeWEF 1.2 (Herdecker Wärmeempfindungs-Fragebogen) overall warmth perception questionnaire

SECONDARY OUTCOMES:
Core body temperature | Baseline (pre intervention), once per week during intervention, 6 weeks after baseline (post intervention), at six-month follow-up
  Core body temperature measured using an infrared tympanical thermometer as used in clinical routine
Face surface temperature | Baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Surface temperature in the face measured using high-resolution infrared thermography
Feet surface temperature | Baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Surface temperature at the feet measured using high-resolution infrared thermography
Hand surface temperature | Baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Surface temperature on the hands measured using high-resolution infrared thermography
Abdomen surface temperature | Baseline (pre intervention) and after 6 weeks (post intervention)
  Surface temperature at the abdomen measured using high-resolution infrared thermography
24-hour feet surface temperature | Over 24 hours at baseline (pre intervention) and over 24 hours 6 weeks after baseline(post intervention)
  24 hour surface temperature at the feet measured using a surface data-logger (i-Button TM)
24-hour hand surface temperature | Over 24 hours at baseline (pre intervention) and over 24 hours 6 weeks after baseline (post intervention)
  24 hour surface temperature on the hands measured using a surface data-logger (i-Button TM)
24-hour abdomen surface temperature | Over 24 hours at baseline (pre intervention) and over 24 hours 6 weeks after baseline (post intervention)
  24 hour surface temperature at the abdomen measured using a surface data-logger (i-Button TM)
24-hour torso surface temperature | Over 24 hours at baseline (pre intervention) and over 24 hours 6 weeks after baseline (post intervention)
  24 hour surface temperature at the upper torso measured using a surface data-logger (i-Button TM)
Body Mass Index | Baseline (pre intervention),weekly during intervention, 6 weeks after baseline (post intervention) and at six-month follow-up
  Body Mass Index (BMI) Calculated as (Weight in Kg)/〖(Height in m)^2〗
Pulse Transit Time (PTT) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  PTT in ms, measured with the GeTeMed Vitaguard 3100
Perfusion Index (PI) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  PI, measured with the GeTeMed Vitaguard 3100
Peak to Peak Time (PPT) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Peak to Peak Time (PPT, ms) measured with the GeTeMed Vitaguard 3100
SlopeInW1 | Continuously over 15 minutes at baseline (pre intervention) and after 6 weeks (post intervention)
  Measured with the GeTeMed Vitaguard 3100
SlopeInW2 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
SlopeInW3 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
SlopeInW4 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Measured with the GeTeMed Vitaguard 3100
Stiffness Index | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
Reflection Index | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
TimeTX | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  TimeTX in ms (millisecond), measured with the GeTeMed Vitaguard 3100
TimeTY | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  TimeTY in ms, measured with the GeTeMed Vitaguard 3100
QuotTYTX | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Measured with the GeTeMed Vitaguard 3100
AreaAX | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
AreaAY | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
QuotAYAX | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Measured with the GeTeMed Vitaguard 3100
AreaAV | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Measured with the GeTeMed Vitaguard 3100
AreaAW | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
QuotAWAV | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
QuotTVTW | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Measured with the GeTeMed Vitaguard 3100
TimeTV | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  TimeTV in ms, measured with the GeTeMed Vitaguard 3100
TimeTW | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  TimeTW in ms, measured with the GeTeMed Vitaguard 3100
MinT1 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Minimum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the beginning of the second peak
MinT2 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Minimum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the beginning of the second peak
MaxT1 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Maximum of the pulse wave measured with the GeTeMed Vitaguard 3100 at the beginning of the first peak
MaxT2 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Maximum of the pulse wave measured with the GeTeMed Vitaguard 3100 at the beginning of the second peak
QuotHRRespRate | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Quotient of heart and respiratory rates measured with the GeTeMed Vitaguard 3100
Heart rate | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  beats per minute (bpm) measured with the GeTeMed Vitaguard 3100
Respiratory rate | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  measured with the GeTeMed Vitaguard 3100
SDNN (standard deviation of normal to normal) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Standard deviation of normal to normal beats, measured with the GeTeMed Vitaguard 3100
RMSSD (Root mean square of successive differences) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Root mean square of successive differences, measured with the GeTeMed Vitaguard 3100
pNN50 | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Number of pairs of successive heart rate intervals that differ by more than 50 ms
HF (high frequency) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline(post intervention)
  Area under the curve between the frequency of 0.15 to 0.4Hz measured with the GeTeMed Vitaguard 3100
LF (low frequency) | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Area under the curve between the frequency of 0.04 to 0.15Hz measured with the GeTeMed Vitaguard 3100
LF/HF-Ratio | Continuously over 15 minutes at baseline (pre intervention) and 6 weeks after baseline (post intervention)
  Ratio of two bands from frequency domain analysis: LF band (0.04-0.15 Hz), HF band (0.15-0.40 Hz), measured with the GeTeMed Vitaguard 3100
Pittsburgh sleep quality index | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the PSQI (Pittsburgh sleep quality index)
Eating Disorder Inventory -2 | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the EDI-2 (Eating Disorder Inventory)
Eating Disorder Examination- Questionnaire | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the EDE-Q (Eating Disorder Examination)
Becks Depressions Inventar | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the BDI-II (Becks Depression Inventar)
Hospital Anxiety and Depression Scale subscale Anxiety | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Anxiety Sum-Score of the HADS (Hospital Anxiety and Depression scale) ranging from 0-21 with a cutoff at >10 (being evaluated as pathological)
Hospital Anxiety and Depression Scale subscale Depression | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Depression Sum-Score of the HADS (Hospital Anxiety and Depression scale) ranging from 0-21 with a cutoff at >10 (being evaluated as pathological)
Body Image State Scale | Baseline (pre intervention),6 weeks after baseline (post intervention), at six-month follow-up
  Mean of all six item values (range from 0-9) with higher values indicating a positive body image state of the BISS (Body Image State Scale)
Positive And Negative Affect Schedule | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the PANAS-X (Positive and negative affect schedule)
Short Form Health Survey 12 | Baseline (pre intervention), 6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the SF-12 (Short Form 12)
Basler Befindlichkeits Skala | Baseline (pre intervention), once per week during intervention, 6 weeks after baseline(post intervention), at six-month follow-up
  Scores of the BBS (Basler Befindlichkeits Skala =basler mood questionnaire)
Body Shape Questionnaire | Baseline (pre intervention), once per week during intervention,6 weeks after baseline (post intervention), at six-month follow-up
  Scores of the BSQ (Body Shape Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr. med., Principal Investigator — ARCIM Institute
Locations (1):
- ARCIM Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No